CLINICAL TRIAL: NCT05102175
Title: Addressing Health Disparities in African Americans - Exploring Sleep and Developing Interventions
Acronym: HD-SLEEP1
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Prachi Singh, Associate Professor, Sleep and Cardiometabolic Health, Pennington Biomedical Research Center
Other Study IDs: PBRC 2020-020-1; U54GM104940 (NIH)
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Sleep
Keywords: African American; Sleep; Research Participation
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- African American adults with poor sleep: Individuals with self-identified poor sleep quality and/or quantity
  Interventions: Other: Focus Group

INTERVENTIONS:
Other: Focus Group — Eligible participants will be invited to a semi-structured focus group discussion. Each group will include 8 -12 participants.

SUMMARY:
The purpose of the HD-SLEEP1 study is to help researchers understand what African Americans know and think about sleep. The investigators also want to know how to encourage people to participate in research studies designed to improve sleep.

DETAILED DESCRIPTION:
African Americans (AAs) sleep worse than whites on average, thus contributing to race disparities in major health outcomes. However, contributors to poorer sleep and effective interventions to improve sleep among AAs is lacking due to under-representation of AAs in sleep research. The investigators propose to address this knowledge gap through engagement with the Baton Rouge African American community. The investigators will use focus groups to determine sleep-related perceptions as well as barriers to sleep research recruitment and retention.

In this study, up to 60 African Americans who self-report poor sleep will be invited to participate in focus group discussions to understand 1) sleep related perceptions; 2) factors influencing participation; and 3) willingness to undertake study procedures typical of sleep research studies such as increasing sleep duration, diagnosing and treating OSA; along with other routine research procedures including blood draws, caloric restriction, and body composition exams.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African American
* Age range: >18 years (inclusive)
* Sex: Both males and females will be allowed to participate in the study
* Self-perceived poor sleep
* Willing to be audio and video recorded

Exclusion Criteria:

* Unable to provide written informed consent
* Unable to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African Americans residing in Greater Baton Rouge area will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Importance of Sleep | 1 day
  Identify if sleep is considered important for health
Knowledge related to components of good sleep | 1 day
  Identify adequate sleep duration, good sleep quality, and absence of sleep disorders as important.
Perceived advantages related to participating in sleep-related | 1 day
  May improve health and quality of life
Identify what challenges prevents participation in sleep-related research | 1 day
  Willingness to undertake sleep related study procedures and time commitment
Identify facilitators to participation in sleep research | 1 day
  At-home assessments, study location, number of study visits

CONTACTS AND LOCATIONS:
Overall Officials: Prachi Singh, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Recruiting core Pennington, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided